CLINICAL TRIAL: NCT06597162
Title: The Effect of Patient Safety Education Using Problem-Based Learning Approach on Nurses Patient Safety Knowledge Levels and Patient Safety Attitudes
Acronym: Problem-Based
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kıbrıs İlim Üniversitesi (Other)
Responsible Party: Principal Investigator, Arzu Gönel, Specialist Nurse, Kıbrıs İlim Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CSU-SBF-AG-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Problem-Based Learning; Nursing; Patient Safety
Keywords: patient safety,; problem based learning; nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education group (Experimental): For participants in the training group, data will be collected face to face in two stages: the pre-test phase and the post-training post-test phase.
  A survey will be distributed to the control group simultaneously with the training group and will be collected as pre-test and post-test, but no training will be given to the control group. Only after the study ends will educational materials be shared with the control group.
  Interventions: Behavioral: education of patient safety
- Control group (No Intervention): Routine care was given to the control group

INTERVENTIONS:
Behavioral: education of patient safety — For participants in the training group, data will be collected face to face in two stages: the pre-test phase and the post-training post-test phase.
  A survey will be distributed to the control group simultaneously with the training group and will be collected as pre-test and post-test, but no training will be given to the control group. Only after the study ends will educational materials be shared with the control group.
  Arms: education group

SUMMARY:
This research was planned to reveal and evaluate the effects of the problems experienced in the Turkish Republic of Northern Cyprus Health System, which takes the Republic of Turkey Health System as an example, on patient safety for nurses and to determine the goals that will lead to a solution. As it is known, there are deficiencies in the patient safety training program and legal regulations covering patient safety in healthcare institutions in TRNC. The training program in this research forms the basis for disseminating such training programs in all health institutions operating in TRNC, ensuring patient safety and providing higher quality and safer care.

DETAILED DESCRIPTION:
This research aims to shed light on the literature and the TRNC Health System. It is envisaged that developing and improving patient safety programs in healthcare institutions, supporting the infrastructure system for the use and development of scientific knowledge focused on patient safety, creating appropriate working environments, and correcting the incorrect behavior of healthcare professionals regarding patient safety will contribute to the development of patient safety and facilitate the delivery of quality patient care. This research was planned to determine the effect of the patient safety training program given using the problem-based learning approach on nurses' patient safety knowledge levels and patient safety attitudes.

ELIGIBILITY:
Inclusion Criteria:

Nurse

* Must work as a nurse
* Must not have received this patient safety training before

Exclusion Criteria:

Nurse

* Should not accept to participate in the research voluntarily
* The data collection form must be filled incompletely

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Safety Information Form | 10 week
  The number of questions prepared to determine the level of knowledge about patient safety is 12. 1 of them is open-ended (definition question), 11 of them are closed-ended-multiple choice questions. In multiple choice survey questions, the answer was considered correct when all correct answers in the options were known. 1 point was given for the correct answer to each question. Thus, the lowest score was 0 and the highest score was 12. The mean and standard deviation of knowledge scores are 7.78 ± 1.84, and the median is 8. Accordingly, the knowledge levels of nurses who received 8 points or less were considered "insufficient", and the knowledge levels of nurses who received 9 points or above were considered "adequate"

SECONDARY OUTCOMES:
Patient Safety Attitude Scale | 10 week
  The scale consists of 46 items and 6 sub-dimensions in total (job satisfaction-11 items, teamwork-12 items, safety climate-5 items, management approach-7 items, identifying stress-5 items and working conditions-6 items). The five-point Likert type scale is scored as "5-completely agree, 4-agree, 3-partially agree, 2-disagree, 1-strongly disagree". Some items of the scale (items 21, 36, 37, 38, 39, 40, 41, 42, 43 and 45) are scored negatively. It was determined that the total Cronbach's alpha value of the scale was .93, and the subscale Cronbach's alpha values were .85, .86, .83, .77, .74, and .72.

CONTACTS AND LOCATIONS:
Locations (1):
- Cyprus Science Univercity, Kyrenia, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10649324/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33926438/
- See also: Related Info — https://inter-publishing.com/index.php/IJHSMS/article/view/1263
- See also: Related Info — https://dergipark.org.tr/tr/pub/hacettepesid/issue/48867/622696